CLINICAL TRIAL: NCT04758806
Title: Fecal Microbial Transplantation for Corticosteroids Non-responders and Non-eligible Patients With Severe Alcoholic Hepatitis
Brief Title: Fecal Microbial Transplantation in Severe Alcoholic Hepatitis
Acronym: FMTH7
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other)
Responsible Party: Principal Investigator, Ľubomír Skladaný MD, PhD, Head, Department of Internal Medicine and HEGITO Liver Unit, Principal Investigator, F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 432/2018-IK
Record Dates: First submitted 2021-01-21; First posted 2021-02-17 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcoholic hepatitis; Nonresponders; fecal microbial transplantation
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Intervention Model Description: Eligible for the study are consecutive consenting adult patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal microbial transplantation from unrelated donor (Experimental): Fecal microbial transplant procured (frozen if needed) from healthy unrelated donors is administered via upper GI tract; predefined single dose is repeated at five consecutive days
  Interventions: Biological: Fecal microbial transplantation

INTERVENTIONS:
Biological: Fecal microbial transplantation — Procured faeces procured from unrelated donor

SUMMARY:
1. A subtype of Alcoholic hepatitis (AH), named severe alcoholic hepatitis (SAH) is associated with high short-term mortality (J Hepatol, 2019)
2. The only SAH treatment option - corticosteroids (CS) - are often contraindicated or ineffective (STOPAH Trial)
3. New treatment modalities for remaining patients are much needed
4. Fecal microbial transplantation (FMT) is one of the promising therapies
5. Investigators aimed to see if FMT improves survival in patients admitted with SAH, not responding to-, or non-eligible for CS.

DETAILED DESCRIPTION:
* FMT via upper GI tract is provided to CS non-responders (NR) or non-eligible (NE) adult patients hospitalized with SAH (determined by the Lille-model).
* Modified version of the Sarin FMT protocol is used with microbiota material procured from unrelated healthy donors.

ELIGIBILITY:
Inclusion Criteria:

* consenting, adult
* severe form of acute alcoholic hepatitis (SAH)
* non-responder to corticosteroids according to the Lille model
* patients with SAH not eligible for corticosteroids based on their contraindications

Exclusion Criteria:

* active infection
* presence of untreated large / high-risk / bleeding esophageal varices
* too sick for any therapy / futility (chronic extrahepatic organ failures, no potential for recovery, etc)
* malignancy except for hepatocellular carcinoma in Milan criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28-day
  Overall mortality
Mortality | 90-day
  Overall mortality
Mortality | 1 year
  Overall mortality

SECONDARY OUTCOMES:
Acute on chronic liver failure | In-Hospital
  Acute on chronic liver failure by European definition

CONTACTS AND LOCATIONS:
Overall Officials: Lubomir Skladany, MD, PhD, Principal Investigator — Head Dept Internal Medicine F.D.Roosevelt Teaching Hospital Banska Bystrica Slovakia
Locations (1):
- F.D.Roosevelt Teaching Hospital, Banská Bystrica, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
On request by institution of interest, e.g. on submission to medical journal / by editorial office; by auditing authority
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: First release of results is expected in 2021, final analysis in 2022
Access Criteria: General Data Protection Regulation (GDPR) compliance Editorial office approved member Auditing authority Authors, meta analysis / systematic review
URL: http://www.fnspfdr.sk